CLINICAL TRIAL: NCT01128764
Title: Integrated Treatment for Comorbid Depression and Obesity in Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Anthony Spirito, Professor, National Institute of Mental Health (NIMH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH083092 (NIH); R34MH083092 (NIH)
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Depression; Overweight
MeSH Terms: conditions — Depression; Overweight | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT for depression and healthy lifestyle plus exercise (Experimental): CBT treatment for depressed teens will be adapted into one integrated protocol that addresses depression using CBT techniques, an exercise component, and advice regarding healthy eating.
  Interventions: Behavioral: CBT for depression and healthy lifestyle plus exercise
- CBT for depression (Active Comparator): CBT for depression only
  Interventions: Behavioral: CBT for depression

INTERVENTIONS:
Behavioral: CBT for depression and healthy lifestyle plus exercise — CBT treatment for depressed teens will be adapted into one integrated protocol that addresses depression using CBT techniques, an exercise component, and advice regarding healthy eating.
  Arms: CBT for depression and healthy lifestyle plus exercise
Behavioral: CBT for depression — Standard CBT treatment for depressed teens that addresses depression using CBT techniques only
  Arms: CBT for depression

SUMMARY:
Lifetime prevalence of major depression is estimated at 28% by age 18 (Lewinsohn et al., 1999), with higher cumulative rates in females (35%) than males (19%). Approximately 17% of children and adolescents in the United States are obese as defined by a BMI above the 95th percentile, with more than 30% falling between the 85th and 95th percentiles (Ogden et al., 2008). Overweight children and adolescents are at increased risk for type 2 diabetes (Pinhas-Hamiel et al., 1996) and overwhelming risk for adult obesity (Guo et al., 1994). There is a substantial percentage of adolescents who are both overweight and depressed with estimates from clinical samples averaging 25%. Treatment of teens with comorbid medical and psychiatric conditions such as overweight/obesity and depression has received little to no attention in the psychosocial treatment research literature. Due to the large number of adolescents who are both depressed and overweight, developing a behavioral treatment that addresses both problems simultaneously has important public health significance. The purpose of this proposal is to combine treatments for depression and overweight to address these co-occurring conditions in one intervention. The long-term objectives of this research are to develop efficient and effective treatments for co-occurring physical and emotional disorders. The research program will be divided into 3 major phases: a development phase (Stage 1a), a pilot study phase (Stage 1b), and a revision phase. During the development phase (Stage 1a), a treatment for overweight teens and CBT treatment for depressed teens will be adapted into one integrated protocol that addresses depression using CBT techniques, an exercise component, and advice regarding healthy eating. As part of this phase, we will adapt existing intervention manuals and therapist training materials, and gain some initial clinical experience with the intervention via an open trial with 6 teens. During the randomized pilot study phase (Stage 1b), the integrated intervention will be compared to a control group receiving CBT treatment for depression alone (N=40 in total). During the pilot phase, the feasibility and acceptability of administering the program will be assessed. In addition, we will compare change in depressed mood at end of treatment and 6 month follow-up periods across the two groups. During the revision phase, the intervention manual will be further developed and refined, based on experiences and observations made during the development and pilot study phases.

ELIGIBILITY:
Inclusion Criteria:

Adolescents must: 1) be between the ages of 12 and 18 years (18 year olds must still be in high school and living at home); 2) be at or above the 85th percentile with reference to age and gender-specific Body Mass Index (BMI); 3) have at least one parent available to participate in the treatment protocol; 4) speak English; 5) agree to study participation and random assignment; and 6) be available for follow-up. In order to meet the depressed mood criterion, adolescents must have a primary diagnosis of major depressive disorder (single or recurrent), based on the KSADS-PL with a CGI-Severity ≥ 3 for depression and CDRS ≥ 36. Participants must be healthy, as established by their primary care physician, in order to participate in the exercise program -

Exclusion Criteria:

Adolescents will be excluded if: 1) they are currently receiving psychotherapy or participating in another weight loss program (only can have been in a weight loss program in the past); 2) they have a medical condition that would interfere with the prescribed dietary plan or participation in physical activity; 3) they are developmentally delayed such that the intervention materials will not be appropriate; 4) they are actively suicidal at intake; 5) they have not been on a stable dose of a psychostimulant for 6 months to ensure that a recently prescribed psychostimulant is not contributing to weight loss; 6) teens on an SSRI will not be allowed to participate due to potential effects of medication on weight loss; 7) they have a substance abuse or dependence diagnosis; or 8) they have failed a medication or psychotherapy trial for depression in the past.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2009-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
depressed mood | baseline, posttreatment , 6 month follow-up

SECONDARY OUTCOMES:
weight | baseline, posttreatment, 6 month foll-up

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Spirito, PhD, Principal Investigator — Brown University; Elissa Jelalian, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Jelalian E, Jandasek B, Wolff JC, Seaboyer LM, Jones RN, Spirito A. Cognitive-Behavioral Therapy Plus Healthy Lifestyle Enhancement for Depressed, Overweight/Obese Adolescents: Results of a Pilot Trial. J Clin Child Adolesc Psychol. 2019;48(sup1):S24-S33. doi: 10.1080/15374416.2016.1163705. Epub 2016 Jun 16. PMID 27310418